CLINICAL TRIAL: NCT03497533
Title: TriCAR-T-CD19 Adoptive Immunotherapy for CD19-positive Refractory/Relapsed Non-Hodgkin Lymphoma
Brief Title: Treatment of Refractory/Relapsed Non-Hodgkin Lymphoma With TriCAR-T_CD19
Acronym: Trident19-H
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Timmune Biotech Inc. (Industry)
Collaborators: Hunan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChiCTR1800014528
Record Dates: First submitted 2018-02-11; First posted 2018-04-13 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Non-hodgkin Lymphoma,B Cell
Keywords: CD19; CAR-T; TriCAR-T-CD19; non-Hodgkin lymphoma; NHL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TriCAR-T-CD19 (Experimental): Tri-functional anti-CD19 chimeric antigen receptor transduced autologous T cells will be administered intravenously
  Interventions: Biological: TriCAR-T-CD19

INTERVENTIONS:
Biological: TriCAR-T-CD19 — A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by a single infusion of CAR transduced autologous T cells administered intravenously at a target dose of 0.5-1 x 10^6 CAR+ T cells/kg

SUMMARY:
This is a single arm, open-label, single-center, phase 1/2 study, to determine the safety and efficacy of TriCAR-T-CD19, an autologous tri-functional anti-CD19 chimeric antigen receptor (CAR)-positive T cell therapy, in refractory/Relapsed Non-Hodgkin Lymphoma (NHL).

DETAILED DESCRIPTION:
The tri-functional anti-CD19 chimeric antigen receptor contains an anti-CD19 scFv, a PD-L1 blocker, and a cytokine complex, enabling the TriCAR-T-CD19 to simultaneously targeting the CD19 positive NHL，blocking the inhibitory PD-L1 signal and stimulating T/NK cell activation and expansion.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects must personally sign and date the consent form before initiating any study specific procedures or activities;
2. All subjects must be able to comply with all the scheduled procedures in the study;
3. Histologically or cytologically confirmed CD19 positive non-Hodgkin lymphoma;
4. Chemotherapy-refractory disease, defined as one or more of the following: Relapsed in 6 months after most recent therapy; Progressive disease in the standard R-CHOP or CHOP chemotherapy; Disease progression or relapsed in ≤12 months of ASCT (must have biopsy proven recurrence in relapsed subjects); If salvage therapy is given post-ASCT, the subject must have had no response to or relapsed after the last line of therapy.
5. No available standard therapy;
6. At least one measurable lesion per revised IWG Response Criteria;
7. Aged 18 to 68 years;
8. Expected survival ≥12 weeks;
9. Eastern cooperative oncology group (ECOG) performance status of ≤2;
10. Systematic usage of immunosuppressive drug or corticosteroid must have been stopped for more than 4 weeks;
11. All other treatment induced adverse events must have been resolved to ≤grade 1;
12. Laboratory tests must fulfill the following criteria: ANC ≥ 1000/uL, HGB >70g/L, Platelet count ≥ 50,000/uL, Creatinine clearance ≤1.5 ULN, Serum ALT/AST ≤2.5 ULN, Total bilirubin ≤1.5 ULN (except in subjects with Gilbert's syndrome);
13. Female must be not pregnant during the study.

Exclusion Criteria:

1. History of malignancy other than nonmelanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast) or follicular lymphoma unless disease free for at least 3 years;
2. History of allogeneic stem cell transplantation;
3. Prior other CAR therapy or other genetically modified T cell therapy;
4. Presence of fungal, bacterial, viral, or other infection that is uncontrolled or requiring IV antimicrobials for management. Simple UTI and uncomplicated bacterial pharyngitis are permitted if responding to active treatment;
5. Subjects with detectable cerebrospinal fluid malignant cells, or brain metastases, or with a history of CNS lymphoma, cerebrospinal fluid malignant cells or brain metastases;
6. Lactating women;
7. Active infection with hepatitis B (HBsAG positive) or hepatitis C virus (anti-HCV positive);
8. Subjects need systematic usage of corticosteroid;
9. History of any gene therapy;
10. Subjects need systematic usage of immunosuppressive drug;
11. Known history of infection with HIV;
12. Planed operation, history of other related disease, or any other related laboratory tests restrict patients for the study;
13. Other reasons the investigator think the patient may not be suitable for the study.

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2018-08-03 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety (Incidence of treatment-related adverse events as assessed by CTCAE v4.0) | 30 Days
  Incidence of treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Complete response rate[CR] (Complete response rate per the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma) | 12 months
  Complete response rate per the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma
Partial response rate [PR] (Partial response rate per the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma) | 12 months
  Partial response rate per the revised International Working Group (IWG) Response Criteria for Malignant Lymphoma
Duration of Response （The time from response to relapse or progression） | 12 months
  The time from response to relapse or progression
Progression Free Survival（The time from the first day of treatment to the date on which disease progresses.） | 12 months
  The time from the first day of treatment to the date on which disease progresses.
Overall Survival（The number of patient alive, with or without signs of cancer） | 24 months
  The number of patient alive, with or without signs of cancer

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhou, Principal Investigator — Hunan Provincial People's Hospital
Locations (1):
- Hunan Provincial People's Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kalos M, Levine BL, Porter DL, Katz S, Grupp SA, Bagg A, June CH. T cells with chimeric antigen receptors have potent antitumor effects and can establish memory in patients with advanced leukemia. Sci Transl Med. 2011 Aug 10;3(95):95ra73. doi: 10.1126/scitranslmed.3002842. PMID 21832238
- [Result] Locke FL, Neelapu SS, Bartlett NL, Siddiqi T, Chavez JC, Hosing CM, Ghobadi A, Budde LE, Bot A, Rossi JM, Jiang Y, Xue AX, Elias M, Aycock J, Wiezorek J, Go WY. Phase 1 Results of ZUMA-1: A Multicenter Study of KTE-C19 Anti-CD19 CAR T Cell Therapy in Refractory Aggressive Lymphoma. Mol Ther. 2017 Jan 4;25(1):285-295. doi: 10.1016/j.ymthe.2016.10.020. Epub 2017 Jan 4. PMID 28129122
- [Result] Neelapu SS, Tummala S, Kebriaei P, Wierda W, Gutierrez C, Locke FL, Komanduri KV, Lin Y, Jain N, Daver N, Westin J, Gulbis AM, Loghin ME, de Groot JF, Adkins S, Davis SE, Rezvani K, Hwu P, Shpall EJ. Chimeric antigen receptor T-cell therapy - assessment and management of toxicities. Nat Rev Clin Oncol. 2018 Jan;15(1):47-62. doi: 10.1038/nrclinonc.2017.148. Epub 2017 Sep 19. PMID 28925994